CLINICAL TRIAL: NCT05537168
Title: Use of Deep Neural Networks and Bayesian Analysis to Identify Risk Factors for Poor Outcome After Pediatric Cardiac Surgery
Brief Title: Bayesian Networks in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, Département of Anesthesiology, Brugmann University Hospital
Other Study IDs: PED_CARDIAC_surg_Bayesian
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cardiac Surgical Procedures; Pediatrics; Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric cardiac surgery: All patients with pediatric cardiac surgery under cardiopulmonary bypass between 2008 and 2018 will be included
  Interventions: Procedure: Pediatric cardiac surgery under cardiopulmonary bypass

INTERVENTIONS:
Procedure: Pediatric cardiac surgery under cardiopulmonary bypass — All patients with pediatric cardiac surgery under cardiopulmonary bypass between 2008 and 2018 operated at our institution

SUMMARY:
Pediatric cardiac surgery with cardiopulmonary bypass is associated with significant morbidity and mortality. Also score systems for risk factors, such as Risk Adjustment for Congenital Heart surgery (RACHS 1) score or the ARISTOTLE score, have been developed, outcome prediction remains difficult. New mathematical methods using deep neural networks associated with Bayesian statistical methods have been developed to give a better understanding of the complex interaction between different risk factors, to identify risk factors and group them in related families. This method has been successfully used to predict mortality in dialysis patient as well as to better describe complex psychiatric syndromes.

The primary hypothesis of this study is that the use of these tools will give a better understanding on the factors affecting outcome after pediatric cardiac surgery.

A network analysis using Gaussian Graphical Models, Mixed Graphical models and Bayesian networks will be used to identify single or groups of risk factors for morbidity and mortality after pediatric cardiac surgery under cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 16 years
* cardiac surgery under cardiopulmonary bypass

Exclusion Criteria:

* ASA (American Society of Anesthesiologists) status 5
* Jehovah's Witness

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients with pediatric cardiac surgery under cardiopulmonary bypass between 2008 and 2018 at our institution
Sampling Method: Non-Probability Sample
Enrollment: 1364 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Outcome predictors | 28 days
  All preoperative, peroperative and postoperative variables will be entered into a deep neural network with Bayesian statistics to identify groups or individual risk factors for postoperative morbidity and mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenkins KJ, Gauvreau K, Newburger JW, Spray TL, Moller JH, Iezzoni LI. Consensus-based method for risk adjustment for surgery for congenital heart disease. J Thorac Cardiovasc Surg. 2002 Jan;123(1):110-8. doi: 10.1067/mtc.2002.119064. PMID 11782764
- [Background] Lacour-Gayet F, Clarke D, Jacobs J, Comas J, Daebritz S, Daenen W, Gaynor W, Hamilton L, Jacobs M, Maruszsewski B, Pozzi M, Spray T, Stellin G, Tchervenkov C, Mavroudis And C; Aristotle Committee. The Aristotle score: a complexity-adjusted method to evaluate surgical results. Eur J Cardiothorac Surg. 2004 Jun;25(6):911-24. doi: 10.1016/j.ejcts.2004.03.027. PMID 15144988
- [Background] Siga MM, Ducher M, Florens N, Roth H, Mahloul N, Fouque D, Fauvel JP. Prediction of all-cause mortality in haemodialysis patients using a Bayesian network. Nephrol Dial Transplant. 2020 Aug 1;35(8):1420-1425. doi: 10.1093/ndt/gfz295. PMID 32040147
- [Background] Till AC, Florquin R, Delhaye M, Kornreich C, Williams DR, Briganti G. A network perspective on abnormal child behavior in primary school students. Psychol Rep. 2023 Aug;126(4):1933-1953. doi: 10.1177/00332941221077907. Epub 2022 Mar 24. PMID 35331028
- [Background] Briganti G, Linkowski P. Item and domain network structures of the Resilience Scale for Adults in 675 university students. Epidemiol Psychiatr Sci. 2019 Apr 22;29:e33. doi: 10.1017/S2045796019000222. PMID 31006419
- [Derived] Florquin R, Florquin R, Schmartz D, Dony P, Briganti G. Pediatric cardiac surgery: machine learning models for postoperative complication prediction. J Anesth. 2024 Dec;38(6):747-755. doi: 10.1007/s00540-024-03377-7. Epub 2024 Jul 19. PMID 39028323